CLINICAL TRIAL: NCT02090764
Title: A Phase III 2 Arms, Multicenter, Randomised, Double-blind Study to Assess the Efficacy and Safety of Ozenoxacin 1% Cream Applied Twice Daily for 5 Days Versus Placebo in the Treatment of Patients With Impetigo
Brief Title: Efficacy and Safety of Ozenoxacin 1% Cream Versus Placebo in the Treatment of Patients With Impetigo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-110881-01
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2016-06

CONDITIONS: Impetigo
MeSH Terms: conditions — Impetigo | interventions — ozenoxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ozenoxacin (Experimental): ozenoxacin cream 1%
  Interventions: Drug: Ozenoxacin
- Placebo (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozenoxacin
  Arms: Ozenoxacin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is multicenter, randomised, placebo controlled, parallel, double blinded , superiority clinical study comparing ozenoxacin cream versus placebo, in patients with a clinical diagnosis of non-bullous or bullous impetigo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bullous or non bullous impetigo. The patient has a total affected area comprised between 1-100 cm2 with surrounding erythema not extending more than 2 cm from the edge of any affected area. In case of multiple affected areas the total area will be the sum of each affected area and will not exceed 100 cm2. Additionally for patients < 12 years the total area will not exceed a maximum of 2% of the body surface area.
* Total Skin Infection Rating Scale (SIRS) score of at least 3, including pus/exudate score of at least 1

Exclusion Criteria:

* Has a bacterial infection, which in the opinion of the investigator, could not be appropriately treated by a topical antibiotic.
* Has systemic signs and symptoms of infection (e.g. a fever; defined as an axillary temperature over 37.2 °C (99.0 °F)

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Caparra Internal Medicine Center, Río Grande, Puerto Rico

REFERENCES:
- [Derived] Hebert AA, Albareda N, Rosen T, Torrelo A, Grimalt R, Rosenberg N, Zsolt I, Masramon X. Topical Antibacterial Agent for Treatment of Adult and Pediatric Patients With Impetigo: Pooled Analysis of Phase 3 Clinical Trials. J Drugs Dermatol. 2018 Oct 1;17(10):1051-1057. PMID 30365584
- [Derived] Rosen T, Albareda N, Rosenberg N, Alonso FG, Roth S, Zsolt I, Hebert AA. Efficacy and Safety of Ozenoxacin Cream for Treatment of Adult and Pediatric Patients With Impetigo: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jul 1;154(7):806-813. doi: 10.1001/jamadermatol.2018.1103. PMID 29898217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 34 sites in Germany, Puerto Rico, Romania, Russia, South Africa, Spain and the United States of America (USA).
Groups:
- Ozenoxacin: ozenoxacin cream 1%
  Ozenoxacin
- Placebo: Placebo cream
  Placebo
Period: Overall Study
Arm/Group | Ozenoxacin | Placebo
Started | 206 | 206
Completed | 200 | 186
Not Completed | 6 | 20
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 0 | 13
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Intercurrent illness and other | 1 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was consider the safety population. Safety population was defined as all patients who received at least one application of study drug.
  One patient was randomised to placebo but never treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ozenoxacin | Placebo | Total
Number analyzed (Participants) | 206 | 205 | 411
Age, Customized [Number; unit: participants]
  >=18 years | 69 | 70 | 139
  >=12 years to <18 years | 23 | 23 | 46
  >= 2 months to <12 years | 114 | 112 | 226
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 107 | 201
  Male | 112 | 98 | 210
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 122 | 139 | 261
  Black | 53 | 38 | 91
  Asian | 16 | 15 | 31
  Mixed Race | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 23 | 23 | 46
  Germany | 21 | 16 | 37
  Romania | 26 | 26 | 52
  Russian Federation | 27 | 30 | 57
  South Africa | 43 | 34 | 77
  Spain | 1 | 2 | 3
  United States | 65 | 74 | 139

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Clinical response (clinical success or clinical failure) at end of therapy (Visit 3) in the intent to treat clinical (ITTC) population.
  Clinical success at V3 was defined as: SIRS score 0 for blistering, exudates/pus, crusting and itching/pain and no more than 1 for erythema/inflammation such that no additional antimicrobial therapy in the baseline (Visit 1) affected area is necessary.
  The skin infection rating scale (SIRS) is a severity index based on five signs or symptoms: blistering, exudate/pus, crusting, erythema/inflammation, itching/pain.
Time Frame: Visit 3 (Day 6-7)
Population: Intent-to-treat clinical (ITTC) population was defined as all randomized patients.
  The % of clinical success for the treatment comparison were calculated excluding the unable to determine: OZN (112/203), PLB (78/199)
Measure: Number; unit: percentage of Participants
Arm/Group | Ozenoxacin | Placebo
Number analyzed (Participants) | 203 | 199
percentage of Participants | 55.2 | 39.2
Statistical Analysis 1: Comparison: Ozenoxacin vs Placebo; The treatment comparison was done using only the outcomes of Clinical success and Clinical failure. The p value of the chi square test (without continuity correction) was provided. The analysis was performed to test the superiority of ozenoxacin versus placebo; Test type: Superiority or Other; p = 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: AEs were elicited from signing the informed consent to the completion of the clinical study (including the Follow up Visit) or premature patient withdrawal from the study. (10-13 days)
Description: The safety population was defined as all patients who recieved at least one application of study drug. One patient was randomised to placebo but never received any treatment.Tthat is why there are only 205 patienst in the placebo group in the safety population.
Arm/Group | Ozenoxacin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/205
Other Adverse Events (participants affected / at risk) | 0/206 | 0/205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any and all data resulting from the Study will not be presented or published in any form or media by the Institution, Investigator or Research Staff without the prior written consent of Sponsor which consent maybe as directed within the Protocol.